CLINICAL TRIAL: NCT01411436
Title: Special Drug Use Investigation of Nexavar (Unresectable Hepatocellular Carcinoma)
Brief Title: Nexavar Post-marketing Surveillance for Hepatocellular Carcinoma in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15039; NEXAVAR-HCC-01 (Other: Company Internal)
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Nexavar; unresectable hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Patients who have received Nexavar for unresectable HCC

SUMMARY:
This study is a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Nexavar for unresectable hepatocellular carcinoma (HCC). The objective of this study is to assess safety and effectiveness of Nexavar under real-life practice conditions. This study is an all case investigation of which the enrollment period is 2 or 3 months (dependent on sites) for Child-Pugh A; for Child-Pugh B or C, the enrollment continues until agreement to stop with Pharmaceuticals Medical Devices Agency (PMDA). All patients who have received Nexavar will be recruited and followed one year since starting Nexavar administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received Nexavar for unresectable hepatocellular carcinoma

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is patients who received Nexavar for unresectable HCC.
Sampling Method: Non-Probability Sample
Enrollment: 1637 (Actual)
Dates: Start 2009-05; Primary Completion 2014-03 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions and serious adverse events in subjects who received Nexavar | After Nexavar administration, up to 1 year

SECONDARY OUTCOMES:
Demography | Baseline
Effectiveness evaluation assessment [overall survival, complete response rate, partial response rate, stable disease rate] by the Response Evaluation Criteria in Solid Tumor (RECIST) | After Nexavar administration, up to 1 year
Effectiveness evaluation assessment [time to progression, response rate, stable disease rate, progression rate] by investigator-determined overall best response | After Nexavar administration, up to 1 year
The status of therapy with Nexavar [duration of treatment, daily dose] in a various settings according to baseline data [such as demographic data, Child-Pugh status, ECOG-PS] | After Nexavar administration, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan

REFERENCES:
- [Derived] Kaneko S, Ikeda K, Matsuzaki Y, Furuse J, Minami H, Okayama Y, Sunaya T, Ito Y, Inuyama L, Okita K. Safety and effectiveness of sorafenib in Japanese patients with hepatocellular carcinoma in daily medical practice: interim analysis of a prospective postmarketing all-patient surveillance study. J Gastroenterol. 2016 Oct;51(10):1011-21. doi: 10.1007/s00535-016-1173-5. Epub 2016 Mar 1. PMID 26931117